CLINICAL TRIAL: NCT03234127
Title: Study of cardiovAscular Contrasted Phenotypes in Patients With FamIliaI hypercholesteRolemia
Acronym: SAFIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC17_0244
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — Whole Genome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atherosclerosis- resistance (Other): FH Patient without atherosclerosis
  Interventions: Genetic: Whole Genome Sequencing
- Control (Other): FH patient with atheroclerosis
  Interventions: Genetic: Whole Genome Sequencing
- the related population without familial hypercholesterolemia (Other): No FH patient
  Interventions: Genetic: Whole Genome Sequencing

INTERVENTIONS:
Genetic: Whole Genome Sequencing — Whole Genome Sequencing Biomarkers analyses
  Other Names: Biological analyzes

SUMMARY:
The main objective of SAFIR is to identify the atherosclerotic genetic factors in these patients, which will identify new therapeutic targets for the treatment of CV and Familial Hypercholesterolemia diseases. In addition, SAFIR will allow the identification of new CV protection biomarkers, which will be useful tools for the development of a personalized medicine for the management of dyslipidemias.

DETAILED DESCRIPTION:
The objective of the SAFIR study is to perform non-invasive coronary vascular phenotyping of familial hypercholesterolemia (FH) families by performing a coronary calcium score and then to detect protective genetic factors in patients who do not have a significant atheroma despite a perturbed biological phenotype.

The investigators will also conduct biochemical, lipidemic and metabolomic analyzes to identify a signature of biomarkers protective of cardiovascular risk in FH patients.

The investigators will use the French FH register, which already includes 3889 patients, to identify these "protected" FH families within the main reference centers for the management of FH for inclusion and follow-up of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient agreeing to sign the consent of the study and the consent of biocollection
* Patient suffering from a familial hypercholesterolemia with a clinically-biologic score DLCN (Dutch Lipid Clinic Network, Annex 2)> 8 and / or a causative mutation identified in the LDL receptor genes, apolipoprotein B100 or Of PCSK9.
* Men ≥ 40 years of age; Female ≥ 50 years
* Patient affiliated to an existing social insurance

The inclusion criteria to be met in the population with known coronary atheroma:

* Subject in secondary prevention of an atheromatous disease: coronary event or ischemic heart disease, irrespective of the result of the coronary calcium score; Ischemic stroke with proven carotid atheromatosis; revascularization (angioplasty, bypass surgery) or amputation in PAD
* Primary prevention topic CV with calcium score ≥ 400 Agatston units

Inclusion criteria to be met in the population without cardiovascular risk:

- No cardiovascular event (including MI, coronary revascularization, angina, stroke &, Transiant ischemic attack of atheromatous origin, PAD) with: For women between 50 and 65 years, a nil calcium score * For women between 65 and 75 years of age, a calcium score** ≤ 10 Agatston units For women over 75 years of age, a calcium score** ≤ 20 Agatston units For men between 40 and 55 years of age, a nil calcium score* for men For men between 55 and 70 years of age, a calcium score** ≤ 10 Agatston units For men over 70 years of age, a calcium score** ≤ 20 Agatston units

* 40 year old men and 50 year old women: less than 6 months old
* 41 year old men and 51 year old women: under 1 year old
* 42 year old men and 52 year old women: under 2 years old
* 43 year old men and 53 year old women: under 3 years old
* 44 year old men and 54 year old women: under 4 years old

  * Less than 5 years

Inclusion criteria to be met in the related population with familial hypercholesterolemia :

* Patient agreeing to sign the consent of the study and the consent of biocollection
* Patient suffering from a familial hypercholesterolemia with a clinically-biologic score DLCN (Dutch Lipid Clinic Network, Annex 2)> 8 and / or a causative mutation identified in the LDL receptor genes, apolipoprotein B100 or Of PCSK9.
* Men or Female ≥ 30 years
* Patient affiliated to an existing social insurance

Inclusion criteria to be met in the related population without familial hypercholesterolemia :

* Patient agreeing to sign the consent of the study and the consent of biocollection
* Patient not suffering from a familial hypercholesterolemia related to one of the members of the population suffering from familial hypercholesterolemia without cardiovascular risk
* Men or Female ≥ 18 years
* Patient affiliated to an existing social insurance

Exclusion Criteria:

* Subject suffering from active cancer or progressive neoplasia
* Subject treated with recent corticosteroid therapy
* Subjects with unsubstituted or poorly controlled hypothyroidism (TSH> normal)
* Subject receiving immunosuppressive or anti-cancer treatment
* Subject refusing to participate
* Subjects under tutelage, curatorship or a safeguard of justice or without social insurance

The exclusion criterion for all populations except the related population without familial hypercholesterolemia:

- Subject with no "definite" familial hypercholesterolemia according to the DLCN score (≤8), after auction. The purpose of the auction will be to rule on the causal nature of an identified mutation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Identification of genes associated with the resistance to development of coronary atherosclerosis in subjects with heterozygous familial hypercholesterolemia | 3 years
  Identification of functional genetic variants by a Whole Genome Sequencing (WGS) approach in case-control analysis (FH without and with advanced coronary atherosclerosis) and/or family analysis (protected and affected relatives)

SECONDARY OUTCOMES:
Identification of new biochemical, lipidemic, metabolomic and metagenomic biomarkers associated with cardiovascular protection in FH patients. | 3 years
  Lipidic panel, phosphocalcic panel, Ceramides, Alipoproteins, Lp(a), lipidomic, LDL size, Phospholipids, TMAO, Carnitin, Cholin, microbiota, metabolomic, LDL Ox, Sterols, Isoprostan, oxidation, inflammation, cytokins, oxidative stress.
Association of arterial stiffness (reflected by the pulse wave velocity) with the development of coronary atherosclerosis in FH patients | 3 years
  Measurement of arterial stiffness measured by popmeter® (pulse wave velocity)
Association of atherosclerosis of supra-aortic trunks (AST) with the development of coronary atherosclerosis in FH patients | 3 years
  Measurement of ASD through arterial Doppler ultrasonography (Intra-media thickness (IMT), degree of stenosis (ESCT), plaque)
Association of atherosclerosis of the lower limbs with the development of coronary atherosclerosis (PAD) in FH patients | 3 years
  Measurement of lower extremity involvement by arterial doppler ultrasonography
Association between aortic valvular score and development of coronary atherosclerosis in FH patients | 3 years
  Measurement of coronary calcium score and aortic valvular score (optional) by a thoracic CT scan
Association between coronary calcium score and aortic valvular score in HF patients | 3 years
  Measurement of coronary calcium score and aortic valvular score (optional) by a thoracic CT scan

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Le Bocage Hospital, Dijon
  - CHRU de Lille, Lille
  - Louis Pradel Cardiovascular Hospital, Lyon
  - La Conception Hospital, Marseille
  - Nantes University Hospital, Nantes
  - Saint-Antoine Hospital, Paris
  - Pitié-Salpêtrière Hospital, Paris
  - Rennes University Hospital, Rennes
  - Toulouse Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided